CLINICAL TRIAL: NCT03758157
Title: welloStationX Determination of Clinical Accuracy
Brief Title: Clinical Accuracy of the welloStationX
Status: Completed | Type: Observational
Sponsor: Wello Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Wello_X
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Temperature Measurement: Each subject will have his or her temperature measured by both the welloStationX Automated Non-Contact Thermometer and the Welch Allyn SureTemp Oral Thermometer.
  Interventions: Diagnostic Test: welloStationX; Diagnostic Test: SureTemp

INTERVENTIONS:
Diagnostic Test: welloStationX — welloStationX is an automated electronic thermometer using an infrared sensor of the surface of the forehead to measure human body skin temperature to screen for fever.
Diagnostic Test: SureTemp — SureTemp is an oral thermometer to measure human body skin temperature.

SUMMARY:
This study evaluates the clinical accuracy of the welloStationX, an automated non-touch self-service electronic thermometer using an infrared sensor of the surface of the forehead to screen for fever.

DETAILED DESCRIPTION:
Traditionally, body temperature is measured using a contact thermometer placed on the forehead, in the mouth, ear, armpit or rectum. Non-contact thermometers allow a person's temperature to be taken with no contact with the person, reducing the discomfort of having to sit still for several minutes. Additionally, there is no need for disinfection between patients to occur, allowing for easier and faster use when screening large numbers of people.

This study is to evaluate the clinical accuracy of the welloStationX, a non-contact thermometer by comparing its measurements with that of the gold standard Welch Allyn SureTemp oral thermometer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* 5 years and up.
* Signed informed consent form.

Exclusion Criteria:

* Use of medications known to affect body temperature (for example, antipyretics, barbiturates, thyroid preparations, antipsychotics, etc.) within 3 hours of the test.
* immunization within seven days of the test

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected from amongst non-profit clinical sites and through social media posts for subjects to come to a test site or to be evaluated in his or her own home in the widespread Dallas/Fort Worth area.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Heller, Study Chair — Wello Inc.
Locations (1):
- Agape Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- welloStationX Automated Non-Contact Thermometer: welloStationX: welloStationX is an automated electronic thermometer using an infrared sensor of the surface of the forehead to measure human body skin temperature to screen for fever.
Period: Overall Study
Arm/Group | welloStationX Automated Non-Contact Thermometer
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temperature Measurement
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.78 (16.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110
febrility [Count of Participants; unit: Participants]
  febrile subjects (temperature >=99.5 deg. C) | 33
  afebrile subjects (temperature < 99.5 deg. C) | 77

OUTCOME MEASURES:

1. Primary Outcome: Clinical Agreement Through Clinical Bias Evaluation
Description: Agreement through clinical bias evaluation was calculated as the Mean Bias ± Standard Deviation (SD) by subtracting the first output measurement recorded with the welloStationX thermometer (DUT) from the corresponding output measurement recorded with the Welch Allyn SureTemp oral thermometer for each subject, and then calculating the Mean Bias ± SD of the biases.
Time Frame: one day
Measure: Mean (Standard Deviation); unit: degrees Farehheit
Arm/Group | Temperature Measurement
Number analyzed (Participants) | 110
degrees Farehheit | 0.04 (0.42)

2. Secondary Outcome: Clinical Repeatability
Description: Clinical Repeatability was calculated using the pooled standard deviations of the triplicate measurements recorded by the welloStationX.
Time Frame: one day
Measure: Number; unit: degrees Farehheit
Arm/Group | Temperature Measurement
Number analyzed (Participants) | 110
degrees Farehheit | 0.062

ADVERSE EVENTS:
Time Frame: One day.
Arm/Group | Temperature Measurement
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03758157/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03758157/SAP_001.pdf